CLINICAL TRIAL: NCT02136069
Title: Phase III, Randomized, Multicenter Double-Blind, Double Dummy Study to Evaluate the Efficacy and Safety of Etrolizumab Compared With Infliximab in Patients With Moderate to Severe Active Ulcerative Colitis Who Are Naive to TNF Inhibitors
Brief Title: A Study Comparing the Efficacy and Safety of Etrolizumab to Infliximab in Participants With Moderate to Severe Ulcerative Colitis Who Are Naïve to Tumor Necrosis Factor (TNF) Inhibitors
Acronym: GARDENIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA29103; 2013-004282-14 (EudraCT Number)
Record Dates: First submitted 2014-04-15; First posted 2014-05-12 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrolizumab; Infliximab; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etrolizumab + Placebo (IV) (Experimental): Participants will receive ertolizumab (SC) Q4W until Week 52 along with placebo matched to infliximab as IV infusion until Week 46.
  Interventions: Drug: Etrolizumab; Other: Placebo (IV)
- Infliximab + Placebo (Injection) (Active Comparator): Participants will receive IV infusion of infliximab at Weeks 0,2, and 6, then every 8 weeks until Week 46 partnered with placebo matched to etrolizumab by SC injection Q4W until Week 52.
  Interventions: Drug: Infliximab; Other: Placebo (Injection)

INTERVENTIONS:
Drug: Etrolizumab — 105 mg administered by subcutaneous (SC) injection once every 4 weeks (Q4W) until Week 52.
  Other Names: PRO145223; RO5490261; RG7413
  Arms: Etrolizumab + Placebo (IV)
Drug: Infliximab — 5 mg/kg of infliximab will be administered by intravenous (IV) infusion at Weeks 0, 2, and 6 and then every 8 weeks until Week 46.
  Arms: Infliximab + Placebo (Injection)
Other: Placebo (IV) — Administered by (IV) infusion at Weeks 0, 2, and 6 and then every 8 weeks until Week 46.
  Arms: Etrolizumab + Placebo (IV)
Other: Placebo (Injection) — Administered by SC injection Q4W until Week 52
  Arms: Infliximab + Placebo (Injection)

SUMMARY:
This is a multicenter, Phase III, randomized, double-blind, double-dummy, parallel-group study to evaluate the safety, efficacy, and tolerability of etrolizumab compared with infliximab in treating participants with moderate to severe ulcerative colitis (UC) who are naive to tumor necrosis factor (TNF) inhibitors. Participants will be randomized in a 1:1 ratio to receive either etrolizumab 105 milligrams (mg) by subcutaneous (SC) injection once every 4 weeks (Q4W) + placebo (intravenous [IV] infusion at Weeks 0, 2, and 6, then once every 8 weeks [Q8W]) or infliximab 5 milligrams/kilogram (mg/kg) IV at Weeks 0, 2, and 6, then Q8W) + placebo (SC Q4W). Time on treatment is 54 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Moderately to severely active UC as determined by the Mayo Clinic Score assessment (MCS)
* Naive to treatment with any anti-TNF inhibitor therapy (including TNF inhibitor biosimilars)
* An inadequate response to or intolerance of prior corticosteroid and/or immunosuppressant treatment
* Background regimen for UC may include oral 5-aminosalicylate (5-ASA), oral corticosteroids, budenoside multi-matrix system (MMX), probiotics, azathioprine (AZA), 6-mercaptopurine (6-MP), or methotrexate (MTX) if doses have been stable during the screening period
* Use of highly effective contraception during and at least 24 weeks after the last dose of study drug

Exclusion Criteria:

* A history of or current conditions and diseases affecting the digestive tract, such as indeterminate colitis, suspicion of ischemic, radiation or microscopic colitis, Crohn's disease, fistulas or abdominal abscesses, colonic mucosal dysplasia, intestinal obstruction, toxic megacolon, or unremoved adenomatous colonic polyps
* Prior or planned surgery for UC
* Past or present ileostomy or colostomy
* Have received non-permitted inflammatory bowel disease (IBD) therapies (including natalizumab, vedolizumab, efalizumab, and tofactinib)
* History of moderate or severe allergic or anaphylactic/anaphylactoid reactions to chimeric, human, or humanized antibodies; fusion proteins, or murine proteins; hypersensitivity to etrolizumab or any of its excipients
* Chronic hepatitis B or C infection, Human deficiency virus (HIV) or tuberculosis (active or latent)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2014-12-24 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (119):
- LKH - Universitätsklinikum der PMU Salzburg, Salzburg, Austria
- Belgium (7):
  - GZA Ziekenhuizen - Campus Sint-Vincentius, Antwerp
  - Imeldaziekenhuis, Bonheiden
  - CHU St Pierre (St Pierre), Brussels
  - Universitair Ziekenhuis Brussel; Neurology, Brussels
  - Cliniques Universitaires Saint-Luc; Pharmacy, Brussels
  - UZ Gent, Ghent
  - AZ Sint Elisabeth Herentals, Herentals
- Canada (6):
  - University of Calgary; Heritage Medical Research Clinic, Calgary, Alberta
  - Zeidler Ledcor Centre - University of Alberta; Division of Gasroenterology, Edmonton, Alberta
  - Guelph GI & Surgery Clinic, Guelph, Ontario
  - Centre de santé et de services sociaux Champlain-Charles-Le Moyne, Greenfield Park, Quebec
  - Hôpital Maisonneuve - Rosemont, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Czechia (8):
  - Vojenska nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Oblastni nemocnice Kladno, a.s., nemocnice Stredoces. kraje; Endoskopicke centrum, Kladno
  - Mestska Nemocnice Ostrava, Ostrava
  - Pardubicka krajska nemocnice, a.s., Pardubice
  - ISCARE a.s., Prague
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad Labem, o.z., Ocni oddeleni, Ústí nad Labem
  - Krajska nemocnice T. Bati, a.s., Zlín
- France (8):
  - CHU de Caen - Hopital Cote de Nacre, Caen
  - CHU Tours - Hôpital Trousseau, Chambray-lès-Tours
  - CHU Clermont Ferrand - Hôtel Dieu, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - CHU Hopital Saint Eloi, Montpellier
  - CHU Nice - Hopital de l'Archet 2, Nice
  - Centre Hospitalier Lyon Sud; Service de Gastro-Enterologie, Pierre-Bénite
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (7):
  - Charite Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - DRK Kliniken Berlin Westend, Berlin
  - Krankenhaus Waldfriede e. V., Berlin
  - Universitätsklinikum Koeln, Cologne
  - Universitätsklinikum Freiburg; Innere Medizin I; Hämatologie, Onkologie und Stammzelltransplantation, Freiburg im Breisgau
  - Gastroenterologie Eppendorfer Baum, Hamburg
  - Universitaetsklinikum Schleswig-Holstein, Campus Kiel, Kiel
- Hungary (10):
  - Bekes Megyei Kozponti Korhaz Dr. Rethy Pal Tagkorhaza, Békéscsaba
  - Semmelweis Egyetem, Budapest
  - Eszak-Kozep-budai Centrum, Uj Szent Janos Korhaz es Szakrendelo, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont; Fázis I-es Klinikai Farmakológiai Vizsgálóhely, Budapest
  - Vasutegeszsegugyi Nonprofit KiemeltenKozhasznu Kft, Debrecen
  - Markhot Ferenc Oktato Korhaz es Rendelointezet, Eger
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz; II. Belgyogyaszat, Miskolc
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Israel (2):
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center; Pediatrics B North and Pediatric Endocrinology Unit, Tel Litwinsky
- Italy (13):
  - Azienda Ospedaliero Universitaria di Parma, Parma, Emilia-Romagna
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Asst Fatebenefratelli Sacco (Fatebenefratelli), Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale Niguarda (Grande Ospedale Metropolitano Niguarda), Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli (Presidio Ospedale Sacco), Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano (MI), Lombardy
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese (MI), Lombardy
  - IRCCS Ospedale Casa Sollievo della Soffenza; Stru Comp di Gastroenterologia ed Endoscopia digest, San Giovanni Rotondo, Lombardy
  - Ospedale Mauriziano Umberto I, Turin, Piedmont
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Azienda Ospedaliera Di Padova, Padua, Veneto
- Netherlands (4):
  - Amsterdam UMC Location VUMC, Amsterdam
  - Amsterdam UMC Location AMC, Amsterdam
  - Maastricht University Medical Center, Maastricht
  - Radboudumc, NL -nijmegen
- Akershus universitetssykehus HF, Lørenskog, Norway
- Portugal (2):
  - Hospital de Braga, Braga
  - Hospital da Senhora da Oliveira Guimarães, Guimarães
- Romania (6):
  - S.C MedLife S.A, Bucharest
  - Institutul Clinic Fundeni Bucuresti, Bucharest
  - Centrul Medical Unirea SRL, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Clinic Judetean Mures, Târgu Mureş
  - Centrul de Gastroenterologie Dr. Goldis, Timișoara
- Singapore General Hospital, Singapore, Singapore
- South Africa (3):
  - Netcare Universitas Private Hospital, Bloemfontein
  - Dr MJ Prins Practice, Cape Town
  - Dr Corne Kruger Inc., Cape Town
- South Korea (18):
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeungnam Univ. Hospital, Daegu
  - Korea University Ansan Hospital, Gyeonggi-do
  - CHA Bundang Medical Centre; CHA university, Seongnam
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
  - Ajou University Hospital, Suwon
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (7):
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, LA Coruña
  - Fundacion Hospital de Alcorcon; Servicio de Digestivo, Alcorcón, Madrid
  - Centro Médico Teknon, Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Danderyds Sjukhus AB, Stockholm, Sweden
- Switzerland (2):
  - Inselspital-Universitaetsspital Bern, Bern
  - Universitätsspital Zürich, Zurich
- United Kingdom (12):
  - The Royal Bournemouth Hospital, Bournemouth
  - Addenbrooke's Hospital, Cambridge
  - University Hospital Coventry, Coventry
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - St James University Hospital, Leeds
  - The Royal London Hospital, London
  - St Thomas Hospital, London
  - King's College London, London
  - Fairfield General Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Danese S, Colombel JF, Lukas M, Gisbert JP, D'Haens G, Hayee B, Panaccione R, Kim HS, Reinisch W, Tyrrell H, Oh YS, Tole S, Chai A, Chamberlain-James K, Tang MT, Schreiber S; GARDENIA Study Group. Etrolizumab versus infliximab for the treatment of moderately to severely active ulcerative colitis (GARDENIA): a randomised, double-blind, double-dummy, phase 3 study. Lancet Gastroenterol Hepatol. 2022 Feb;7(2):118-127. doi: 10.1016/S2468-1253(21)00294-6. Epub 2021 Nov 17. PMID 34798038
- [Derived] Sandborn WJ, Vermeire S, Tyrrell H, Hassanali A, Lacey S, Tole S, Tatro AR; Etrolizumab Global Steering Committee. Etrolizumab for the Treatment of Ulcerative Colitis and Crohn's Disease: An Overview of the Phase 3 Clinical Program. Adv Ther. 2020 Jul;37(7):3417-3431. doi: 10.1007/s12325-020-01366-2. Epub 2020 May 22. PMID 32445184

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Started | 199 | 198
Completed | 165 | 170
Not Completed | 34 | 28
Not completed — UC flare-up | 1 | 0
Not completed — Adverse Event | 6 | 8
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 10 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Non-Compliance | 1 | 0
Not completed — Physician Decision | 5 | 4
Not completed — Withdrawal by Subject | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection) | Total
Number analyzed (Participants) | 199 | 198 | 397
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (15.2) | 39.5 (13.4) | 39.8 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 66 | 147
  Male | 118 | 132 | 250
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 39 | 30 | 69
  Black or African American | 1 | 0 | 1
  White | 150 | 158 | 308
  Other | 9 | 10 | 19
Mayo Clinic Score (MCS) ≤9 or ≥10 at Baseline [Count of Participants; unit: Participants] — Measure Description: Participants were stratified by concomitant treatment with corticosteroids (yes/no) at randomization, concomitant treatment with immunosuppressants (yes/no) at randomization, and disease activity measured during screening (MCS ≤9/MCS ≥10). The MCS ranges from 0 to 12 and is a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and physician's global assessment (PGA) subscore. Each of the four assessments was rated with a score from 0 to 3, with higher scores indicating more severe disease. Population: For the Infliximab arm, only 197 subjects had MCS categorical scores available for baseline.
  Participants
    MCS ≤9: number analyzed (Participants) | 199 | 197 | 396
    MCS ≤9 | 139 | 147 | 286
    MCS ≥10: number analyzed (Participants) | 199 | 197 | 396
    MCS ≥10 | 60 | 50 | 110
Baseline Treatment: None, Corticosteroids (CS) or Immunosuppressants (IS) Alone, or Both CS and IS [Count of Participants; unit: Participants] — Participants were stratified by concomitant treatment with corticosteroids (yes/no) at randomization, concomitant treatment with immunosuppressants (yes/no) at randomization, and disease activity measured during screening (MCS ≤9/MCS ≥10).
  Participants
    Corticosteroids (CS) Alone | 59 | 56 | 115
    Immunosuppressants (IS) Alone | 40 | 36 | 76
    Both CS and IS | 25 | 30 | 55
    None | 75 | 76 | 151

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Both Clinical Response at Week 10 and Clinical Remission at Week 54, as Determined by the Mayo Clinic Score (MCS)
Description: Mayo Clinic Score (MCS) is a composite of 4 assessments, each rated from 0-3: stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores indicate more severe disease.
  Clinical Response is MCS with ≥3-point decrease and 30% reduction from baseline as well as ≥1-point decrease in rectal bleeding subscore or an absolute rectal bleeding score of 0 or 1.
  Clinical Remission is MCS ≤2 with individual subscores ≤1.
Time Frame: Week 10, Week 54
Measure: Number; unit: percentage of participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
percentage of participants | 18.6 | 19.7
Statistical Analysis 1: Comparison: Etrolizumab + Placebo (IV) vs Infliximab + Placebo (Injection); Test type: Superiority; p = 0.8114, Cochran-Mantel-Haenszel; Adjusted Difference in Remission Rates = -0.9, 95% CI [-8.70 to 6.83]

2. Secondary Outcome: Percentage of Participants Achieving Clinical Remission at Week 10, Defined as MCS ≤2 With Individual Subscores ≤1
Description: MCS is a composite of 4 assessments, each rated from 0-3: stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores indicate more severe disease.
Time Frame: Week 10
Measure: Number; unit: percentage of participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
percentage of participants | 20.6 | 32.8
Statistical Analysis 1: Comparison: Etrolizumab + Placebo (IV) vs Infliximab + Placebo (Injection); Test type: Non-Inferiority — with margin -12.5%; p = 0.1293, Cochran-Mantel-Haenszel — p-values are not multiplicity adjusted; A Farrington-Manning non-inferiority test was used to determine the nominal p-value; Adjusted Difference in Remission Rates = -12.0, 95% CI 2-sided [-20.50 to -3.26]

3. Secondary Outcome: Percentage of Participants Achieving Clinical Remission at Week 54, as Determined by the MCS
Description: Mayo Clinic Score (MCS) is a composite of 4 assessments, each rated from 0-3: stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores indicate more severe disease.
  Clinical Remission is MCS ≤2 with individual subscores ≤1.
Time Frame: Week 54
Measure: Number; unit: percentage of participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
percentage of participants | 20.1 | 23.7
Statistical Analysis 1: Comparison: Etrolizumab + Placebo (IV) vs Infliximab + Placebo (Injection); Test type: Superiority; p = 0.4056, Cochran-Mantel-Haenszel — p-values are not multiplicity adjusted; Adjusted Difference in Remission Rates = -3.4, 95% CI 2-sided [-11.53 to 4.74]

4. Secondary Outcome: Percentage of Participants Achieving Clinical Remission at Both Week 10 and Week 54, as Determined by the MCS
Description: MCS is a composite of 4 assessments, each rated from 0-3: stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores indicate more severe disease.
  Clinical Remission is MCS ≤2 with individual subscores ≤1.
Time Frame: Week 10 and Week 54
Measure: Number; unit: percentage of participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
percentage of participants | 10.6 | 13.1
Statistical Analysis 1: Comparison: Etrolizumab + Placebo (IV) vs Infliximab + Placebo (Injection); Test type: Superiority; p = 0.4591, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted Difference in Remission Rates = -2.4, 95% CI 2-sided [-8.88 to 4.14]

5. Secondary Outcome: Percentage of Participants Achieving Clinical Remission at Week 54 Among Those With a Clinical Response at Week 10, as Determined by the MCS
Description: MCS is a composite of 4 assessments, each rated from 0-3: stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores indicate more severe disease.
  Clinical Remission is MCS ≤2 with individual subscores ≤1.
  Clinical Response is MCS with ≥3-point decrease and 30% reduction from baseline as well as ≥1-point decrease in rectal bleeding subscore or an absolute rectal bleeding score of 0 or 1.
Time Frame: Week 10 and Week 54
Population: Participants that achieved a Clinical Response at Week 10
Measure: Number; unit: percentage of participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 98 | 117
percentage of participants | 37.8 | 33.3
Statistical Analysis 1: Comparison: Etrolizumab + Placebo (IV) vs Infliximab + Placebo (Injection); Test type: Superiority; p = 0.4196, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted Difference in Remission Rates = 5.3, 95% CI 2-sided [-7.54 to 18.13]

6. Secondary Outcome: Percentage of Participants With Improvement in Endoscopic Appearance of the Mucosa at Week 10, Determined by the MCS
Description: MCS is a composite of 4 assessments, each rated from 0-3: stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores indicate more severe disease.
  Improvement in endoscopic appearance of the mucosa is Endoscopy subscore ≤1.
Time Frame: Baseline to Week 10
Measure: Number; unit: percentage of participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
percentage of participants | 36.7 | 49.5
Statistical Analysis 1: Comparison: Etrolizumab + Placebo (IV) vs Infliximab + Placebo (Injection); Test type: Superiority; p = 0.0118, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted Difference in Response Rates = -12.4, 95% CI 2-sided [-21.84 to -2.66]

7. Secondary Outcome: Percentage of Participants With Improvement in Endoscopic Appearance of the Mucosa at Week 54, as Determined by the MCS
Description: as for outcome 6
Time Frame: Baseline to Week 54
Measure: Number; unit: percentage of participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
percentage of participants | 27.1 | 32.3
Statistical Analysis 1: Comparison: Etrolizumab + Placebo (IV) vs Infliximab + Placebo (Injection); Test type: Superiority; p = 0.2845, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted Difference in Response Rates = -4.9, 95% CI 2-sided [-13.76 to 4.12]

8. Secondary Outcome: Percentage of Participants With Improvement in Endoscopic Appearance of the Mucosa at Both Week 10 and Week 54, as Determined by the MCS
Description: as for outcome 6
Time Frame: Baseline to Week 10, Week 54
Measure: Number; unit: percentage of participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
percentage of participants | 18.1 | 24.7
Statistical Analysis 1: Comparison: Etrolizumab + Placebo (IV) vs Infliximab + Placebo (Injection); Test type: Superiority; p = 0.1234, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted Difference in Response Rates = -6.3, 95% CI 2-sided [-14.30 to 1.84]

9. Secondary Outcome: Percentage of Participants With Endoscopic Remission at Week 54, as Determined by the MCS
Description: MCS is a composite of 4 assessments, each rated from 0-3: stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores indicate more severe disease.
  Endoscopic Remission is Endoscopy subscore = 0.
Time Frame: Week 54
Measure: Number; unit: percentage of participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
percentage of participants | 17.6 | 22.7
Statistical Analysis 1: Comparison: Etrolizumab + Placebo (IV) vs Infliximab + Placebo (Injection); Test type: Superiority; p = 0.2168, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted Difference in Remission Rates = -5.0, 95% CI 2-sided [-12.84 to 2.94]

10. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Week 10, as Determined by the MCS
Description: MCS is a composite of 4 assessments, each rated from 0-3: stool frequency, rectal bleeding, endoscopy, and physician's global assessment. Higher scores indicate more severe disease.
  Clinical Response is MCS with ≥3-point decrease and 30% reduction from baseline as well as ≥1-point decrease in rectal bleeding subscore or an absolute rectal bleeding score of 0 or 1.
Time Frame: Week 10
Measure: Number; unit: percentage of participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
percentage of participants | 49.2 | 59.1
Statistical Analysis 1: Comparison: Etrolizumab + Placebo (IV) vs Infliximab + Placebo (Injection); Test type: Superiority; p = 0.0564, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted Difference in Response Rates = -9.5, 95% CI 2-sided [-19.06 to 0.29]

11. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Both Weeks 10 and 54, as Determined by the MCS
Description: as for outcome 10
Time Frame: Week 10, Week 54
Measure: Number; unit: percentage of participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
percentage of participants | 23.1 | 29.3
Statistical Analysis 1: Comparison: Etrolizumab + Placebo (IV) vs Infliximab + Placebo (Injection); Test type: Superiority; p = 0.1729, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted Difference in Response Rates = -6.0, 95% CI 2-sided [-14.51 to 2.70]

12. Secondary Outcome: Percentage of Participants That Achieve Clinical Remission Corticosteroid-Free at Week 54 (Off Corticosteroid for at Least 24 Weeks Prior to Week 54) Among Those Who Were Receiving Corticosteroids at Baseline, as Determined by the MCS
Description: as for outcome 4
Time Frame: Week 54
Population: Participants that were receiving corticosteroids at baseline
Measure: Number; unit: percentage of participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 84 | 86
percentage of participants | 15.5 | 17.4
Statistical Analysis 1: Comparison: Etrolizumab + Placebo (IV) vs Infliximab + Placebo (Injection); Test type: Superiority; p = 0.8941, Cochran-Mantel-Haenszel — p-value has not been adjusted for multiplicity; Adjusted Difference in Remission Rates = -0.8, 95% CI 2-sided [-12.01 to 10.68]

13. Secondary Outcome: Number of Participants With Adverse Events, Severity Determined According to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI CTCAE v4.0)
Description: All adverse events (AEs) were graded for severity using the NCI-CTCAE v4.0. Any AE not specifically listed was assessed per the following 5 grades: Grade 1 = mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated. Grade 2 = moderate; minimal, local, or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living. Grade 3 = severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living. Grade 4 = life-threatening consequences or urgent intervention indicated. Grade 5 = death related to AE. Not all grades are appropriate for all AEs; some AEs have fewer than 5 options. The terms "severe" and "serious" are not synonymous and are independently assessed for each AE. Multiple occurrences of AEs were counted only once per participant at the highest (worst) grade.
Time Frame: Baseline until the end of study (up to 66 weeks)
Measure: Number; unit: participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
participants
  Grade 1 | 42 | 48
  Grade 2 | 72 | 74
  Grade 3 | 35 | 23
  Grade 4 | 5 | 5
  Grade 5 | 0 | 1

14. Secondary Outcome: Number of Participants With Adverse Events Leading to Study Drug Discontinuation
Time Frame: Baseline until the end of study (up to 66 weeks)
Measure: Number; unit: participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
participants | 29 | 25

15. Secondary Outcome: Number of Participants With Infection-Related Adverse Events, Severity Determined According to the NCI CTCAE v4.0
Description: All AEs were graded for severity using the NCI-CTCAE v4.0. Any AE not specifically listed was assessed per the following 5 grades: Grade 1 = mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated. Grade 2 = moderate; minimal, local, or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living. Grade 3 = severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living. Grade 4 = life-threatening consequences or urgent intervention indicated. Grade 5 = death related to AE. Not all grades are appropriate for all AEs; some AEs have fewer than 5 options. The terms "severe" and "serious" are not synonymous and are independently assessed for each AE. Multiple occurrences of AEs were counted only once per participant at the highest (worst) grade.
Time Frame: Baseline until the end of study (up to 66 weeks)
Measure: Number; unit: participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
participants
  Grade 1 | 28 | 27
  Grade 2 | 31 | 29
  Grade 3 | 8 | 4
  Grade 4 | 2 | 1
  Grade 5 | 0 | 0

16. Secondary Outcome: Number of Participants With Serious Infection-Related Adverse Events
Time Frame: Baseline until the end of study (up to 66 weeks)
Measure: Number; unit: participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
participants | 11 | 3

17. Secondary Outcome: Number of Participants With Malignancies
Time Frame: Baseline until the end of study (up to 66 weeks)
Measure: Number; unit: participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
participants | 3 | 1

18. Secondary Outcome: Number of Participants With Injection-Site Reactions, Severity Determined According to the NCI CTCAE v4.0
Description: as for outcome 13
Time Frame: Baseline until the end of study (up to 66 weeks)
Measure: Number; unit: participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
participants
  Grade 1 | 7 | 5
  Grade 2 | 0 | 2
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

19. Secondary Outcome: Number of Participants With Hypersensitivity Reaction Events, Severity Determined According to the NCI CTCAE v4.0
Description: as for outcome 13
Time Frame: Baseline until the end of study (up to 66 weeks)
Measure: Number; unit: participants
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 199 | 198
participants
  Grade 1 | 0 | 2
  Grade 2 | 0 | 7
  Grade 3 | 0 | 1
  Grade 4 | 0 | 2
  Grade 5 | 0 | 0

20. Secondary Outcome: Pharmacokinetics: Etrolizumab Serum Concentration
Time Frame: Weeks 2, 10, 12, 30, and 54
Population: A subset of etrolizumab-treated participants who received at least one dose of study drug and had at least one quantifiable concentration measured post baseline.
Measure: Mean (Standard Deviation); unit: microgram/milliliter
Arm/Group | Etrolizumab + Placebo (IV)
Number analyzed (Participants) | 153
microgram/milliliter
  Week 2: number analyzed (Participants) | 149
  Week 2 | 7.64 (2.75)
  Week 10: number analyzed (Participants) | 144
  Week 10 | 12.0 (4.63)
  Week 12: number analyzed (Participants) | 111
  Week 12 | 6.92 (3.18)
  Week 32: number analyzed (Participants) | 85
  Week 32 | 13.9 (5.96)
  Week 54: number analyzed (Participants) | 73
  Week 54 | 13.2 (5.68)

21. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Overall Score at Weeks 10, 30, and 54
Description: The IBDQ is used to assess participant's health-related quality of life (QOL). The 32-item questionnaire contains four domains: bowel symptoms (10 items), systemic symptoms (5 items), emotional function (12 items), and social function (5 items). The items are scored on a 7-point Likert scale with a higher score indicating better health-related QOL.
  IBDQ score is a total score summed up from across all 32 questions on the questionnaire. The score can range from 32-224 and the higher score indicates a better quality of life.
Time Frame: Weeks 10, 30, and 54
Population: Participants that completed the IBDQ Questionnaire at baseline and at the respective Time Points
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
Number analyzed (Participants) | 165 | 156
scores on a scale
  Week 10 | 43.2 (36.6) | 45.1 (39.4)
  Week 30: number analyzed (Participants) | 102 | 110
  Week 30 | 53.5 (40.8) | 59.6 (34.4)
  Week 54: number analyzed (Participants) | 82 | 90
  Week 54 | 58.2 (32.9) | 63.2 (38.5)
Statistical Analysis 1: Comparison: Etrolizumab + Placebo (IV) vs Infliximab + Placebo (Injection); Test type: Superiority — Week 10; p = 0.4106, ANCOVA — p-value has not been adjusted for multiplicity; Difference in Adjusted Means = -3.1, 95% CI 2-sided [-10.6 to 4.3]
Statistical Analysis 2: Comparison: Etrolizumab + Placebo (IV) vs Infliximab + Placebo (Injection); Test type: Superiority — Week 30; p = 0.1434, ANCOVA — p-value has not been adjusted for multiplicity; Difference in Adjusted Means = -5.7, 95% CI 2-sided [-13.3 to 1.9]
Statistical Analysis 3: Comparison: Etrolizumab + Placebo (IV) vs Infliximab + Placebo (Injection); Test type: Superiority — Week 54; p = 0.1103, ANCOVA — p-value has not been adjusted for multiplicity; Difference in Adjusted Means = -6.1, 95% CI 2-sided [-13.6 to 1.4]

22. Secondary Outcome: Number of Participants With Anti-Therapeutic Antibodies (ATAs) to Etrolizumab
Time Frame: Weeks 0, 4, 10, 12, 30, and 54
Population: A subset of etrolizumab-treated participants with at least one baseline or post-baseline ATA result from at least one sample.
Measure: Number; unit: participants
Arm/Group | Etrolizumab + Placebo (IV)
Number analyzed (Participants) | 196
participants | 69

ADVERSE EVENTS:
Time Frame: Baseline until the end of study (up to 66 weeks)
Arm/Group | Etrolizumab + Placebo (IV) | Infliximab + Placebo (Injection)
All-Cause Mortality (participants affected / at risk) | 0/199 | 1/198
Serious Adverse Events (participants affected / at risk) | 32/199 | 20/198
Other Adverse Events (participants affected / at risk) | 94/199 | 80/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etrolizumab + Placebo (IV) (N=199) | Infliximab + Placebo (Injection) (N=198)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 12 (12) | 11 (11)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 3 (3) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis listeria (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Stitch abscess (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Central nervous system vasculitis (Nervous system disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etrolizumab + Placebo (IV) (N=199) | Infliximab + Placebo (Injection) (N=198)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 5 (6)
Colitis ulcerative (Gastrointestinal disorders) | 45 (47) | 33 (36)
Diarrhoea (Gastrointestinal disorders) | 11 (12) | 4 (4)
Nausea (Gastrointestinal disorders) | 10 (10) | 4 (4)
Nasopharyngitis (Infections and infestations) | 22 (30) | 23 (30)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (24) | 15 (16)
Headache (Nervous system disorders) | 22 (30) | 19 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT02136069/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT02136069/SAP_001.pdf